CLINICAL TRIAL: NCT00182598
Title: Applying Web Technology to Buprenorphine Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Development and Research Institutes, Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R42DA014727 (NIH)
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2008-08-13 (Estimated); Status verified 2008-08

CONDITIONS: Adult Opioid-Dependence
Keywords: buprenorphine; computer; treatment; opioid; heroin
MeSH Terms: conditions — Opioid-Related Disorders

INTERVENTIONS:
Procedure: computer-based psychoeducational intervention
Procedure: community-based substance abuse counseling

SUMMARY:
The purpose of this clinical trial is to examine the efficacy and cost-effectiveness of an interactive, computer-based psychoeducational system when used by opioid-dependent patients in office-based buprenorphine treatment.

DETAILED DESCRIPTION:
The partial opioid agonist, buprenorphine, was recently approved by the FDA for the treatment of opioid-dependence and will be available via physician prescription, enabling a greatly needed expansion of access to opioid treatment services. However, physicians, because of considerable demands on their time, will likely be unable to provide or coordinate referral for opioid-dependent patients to receive supplemental educational interventions that are critical to the success of their treatment. To address this challenge, we are developing an interactive, web-based patient education system for opioid-dependent individuals in office-based buprenorphine treatment. In this system, we plan to provide patients with educational interventions of demonstrated efficacy (e.g., information about buprenorphine, HIV/AIDS education, relapse prevention skills training). In Phase I, we demonstrated the scientific, technical and commercial merit and feasibility of this web-based patient education system by developing several modules of the program as well as the appropriate technology for the program to be delivered in an office-based setting. We subsequently assessed these modules in the context of feedback sessions conducted with opioid-dependent individuals in a lab designed to mimic the technical constraints of a physician's office. Results demonstrated that this system represents a viable approach to patient education in office-based buprenorphine treatment. During Phase II, we plan to complete our research and development efforts on this project. We will complete all educational modules of the system. We will also develop a "customization program" that patients can use to help them identify the optimal order in which they may access the program modules while in treatment. Additionally, we will establish an electronic reporting system that will provide physicians prescribing buprenorphine with patient activity reports, enabling them to track and document patient progress through the system and ensure that patients are compliant with ancillary educational interventions. Additionally, we plan to conduct a randomized, controlled trial to evaluate the efficacy and cost-effectiveness of this patient education system delivered via the Internet compared to the delivery of patient educational services by community-based treatment facilities outside of the office-based setting. This system will provide patients, physicians and the larger community with assurance that patients in office-based buprenorphine treatment are receiving ancillary services along with their medication, thereby improving their likelihood for a successful treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Opioid dependence
* Adults ( >/= 18 years)
* In first month of office-based buprenorphine maintenance treatment

Exclusion Criteria:

* In buprenorphine-assisted taper

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2004-12

PRIMARY OUTCOMES:
opiate use

SECONDARY OUTCOMES:
treatment retention
other drug use
HIV risk behavior
opiate craving
psychosocial status
feedback on intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Marsch, PhD, Principal Investigator — National Development and Research Institutes, Inc.
Locations (2):
- United States (2):
  - Dr. Steven Lee, New York, New York
  - Dr. Tania Taubes, New York, New York